CLINICAL TRIAL: NCT05003557
Title: Facteurs Pronostiques Des Troubles Fonctionnels Neurologiques : étude rétrospective et évaluation d'un Score
Brief Title: Prognostic Outcome Score in Functional Neurological Disorders
Acronym: POSiF
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC21.167; 2021-A01181-40 (Other: ID RCB)
Record Dates: First submitted 2021-07-06; First posted 2021-08-12 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Functional Neurological Symptom Disorder
Keywords: psychogenic
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire administration — 3 different questionnaires are going to be administered to each participant,
  * concerning the current health situation
  * the SF 36
  * the IPQ-R questionnaire

SUMMARY:
Monocentric retrospective observational cohort study, using a consecutive series of patients hospitalized for FND from 2012 to 2015 in the neurology department A of the Grenoble Alpes University Hospital. During the discharge staff, an estimation of different prognostic factors had been performed in a consensual way by the medical team for all subjects. It is possible to calculate a score (POS) retrospectively from the data collected during the staff. The following items were evaluated on a Likert scale from 1 to 5: quality of adherence to the diagnosis, presence of a current medical treatment, presence of a similar history, duration of evolution of the disorders presented, ability to verbalize, presence of a social adaptation to the disorders, access to psychiatric care.

The aim of the study will be to study the properties of the calculated score according to the evolution of the patients. The investigators will retrospectively collect information from the medical records. In addition, the evolution of the disorder since the initial hospitalization will be analyzed via a self-evaluation by the subjects and the study of the current medical records.

The investigators will also collect information on the quality of life of the patients in the cohort and their perception of the disease at present.

Using a Clinical Global Impression (CGI-I) scale on FNDstatus, subjects will be classified into two groups by the two principal investigators (Dr. Vercueil, M. Bratanov): the first with a favorable evolution (disappearance of symptoms at the last follow-up, low health care consumption, favorable self-assessment of health status, persistence of symptoms at a low level of disability, satisfactory social and professional integration), and the second with an unfavorable evolution (persistence of symptoms at a disabling level, high health care consumption, unfavorable self-assessment of health status, lack of social and professional integration, multiple medical consultations). The prognostic properties of the POS score will be then studied in order to establish an ROC curve that will allow to classify patients in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Male or female gender
* Hospitalization in Neurology Department A from 2012 to 2015 with a final retained diagnosis of NFT
* POS score at time of hospitalization available

Exclusion Criteria:

* Patient under legal protection
* Inability to complete a self-questionnaire
* Minor subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized in neurology ward from 2012 to 2015 and presenting with FND
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Clinical evolution according the Clinical Global Impression scale | continuously through study completion, an average of 1 year
  Using a Clinical Global Impression (CGI-I) scale on FNDstatus, subjects will be classified into two groups by the two principal investigators (Dr. Vercueil, M. Bratanov): the first with a favorable evolution (disappearance of symptoms at the last follow-up, low health care consumption, favorable self-assessment of health status, persistence of symptoms at a low level of disability, satisfactory social and professional integration), and the second with an unfavorable evolution (persistence of symptoms at a disabling level, high health care consumption, unfavorable self-assessment of health status, lack of social and professional integration, multiple medical consultations)

SECONDARY OUTCOMES:
Quality of life of each patient | continuously through study completion, an average of 1 year
  using the 36-Item Short Form Survey (SF-36) Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved.All items are scored so that a high score defines a more favorable health state.
Illness perception as reported by each patient | continuously through study completion, an average of 1 year
  Using the Revised Illness Perception Questionnaire(IPQ-R)
  Coding:
  for identity scale yes = 1; no = 0 for other items: strongly disagree =1, disagree =2, neither agree or disagree = 3, agree = 4, strongly agree = 5
  High scores on the identity, timeline, consequences, and cyclical dimensions represent strongly held beliefs about the number of symptoms attributed to the illness, the chronicity of the condition, the negative consequences of the illness, and the cyclical nature of the condition.
  High scores on the personal control, treatment control and coherence dimensions, represent positive beliefs about the controllability of the illness and a personal understanding of the condition.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Vercueil, MD; PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No